CLINICAL TRIAL: NCT04970745
Title: Application of Tremor Analysis in Parkinson's Disease and Its Related Diseases
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2018222
Record Dates: First submitted 2021-06-27; First posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-06

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- high-risk: After performing midbrain ultrasound and tremor analysis, patients with positive results of both tests are considered very high-risk patients,
  Interventions: Other: Transcranial parenchymal color Doppler ultrasound (TCS); Other: Electromyography (EMG) tremor analysis
- risk: After performing midbrain ultrasound and tremor analysis, patients with positive results of 1 out of 2 tests are considered risk patients
  Interventions: Other: Transcranial parenchymal color Doppler ultrasound (TCS); Other: Electromyography (EMG) tremor analysis
- low-risk: After performing midbrain ultrasound and tremor analysis, patients with negative results of both tests are considered risk patients
  Interventions: Other: Transcranial parenchymal color Doppler ultrasound (TCS); Other: Electromyography (EMG) tremor analysis

INTERVENTIONS:
Other: Transcranial parenchymal color Doppler ultrasound (TCS) — tracing the nigrostriatal echogenic area
Other: Electromyography (EMG) tremor analysis — observed 1, frequency 2, amplitude (amplitude) 3, correlation between the two sides 4, load and post-drug test differences

SUMMARY:
This is a longitudinal study to evaluate the brainstem of patients at different stages through VEMP neck, masticatory muscle and eye tests on patients with early and middle-advanced PD (20 cases each) and healthy controls (40 cases) The function of various parts is affected. At the same time, combining the patient's neurological function score and non-motor symptom score to find evidence of early involvement and early intervention.

DETAILED DESCRIPTION:
[Background] Tremor is an important symptom of extrapyramidal diseases, and it is also an early symptom of a variety of complex diseases. The classification of tremor has not been completely unified, mainly including essential tremor, Parkinson's disease tremor, etc., each form of tremor has Crossover and connection make clinical differential diagnosis difficult. At the same time, many diseases related to tremor lack pathological, serological and imaging characteristic changes. Therefore, it is particularly important to find accurate and objective evaluation indicators for tremor.

By recording a pair of antagonist muscles (active muscles and passive muscles), electromyography can objectively record the type, degree, amplitude, burst pattern (whether the burst activity of the antagonistic muscles are synchronized or alternate), and weight-bearing The effect of drugs on tremor is very valuable for the diagnosis and differential diagnosis of tremor; especially for patients with Parkinson's disease, it can be several years or even decades before they develop motor symptoms, that is, tremor, rigidity, slowness of movement, and postural instability. There are a wide range of non-motor symptoms, such as smell, mood, sleep, mental behavior and many other aspects. Compared with dyskinesia, non-motor symptoms are both a precursor to the onset and an indication of disease progression. Fully understanding and exploring the law of the occurrence and development of these non-motor symptoms can provide clues for our early diagnosis and provide us with opportunities for early implementation of neuroprotective treatment.

The early clinical symptoms of Parkinson's disease (Pakinson's disease, PD) are often atypical, and it is difficult to diagnose it only based on the history and clinical manifestations. However, when the diagnosis is made when the clinical symptoms are obvious, the patient's substantia nigra dopamine neurons have been reduced by 60-70%, and the opportunity for early treatment is lost. A Berg study also showed that treatment when most neurons in the pre-exercise period have not undergone degeneration can better protect the nerves and may delay the clinical progress of PD. Therefore, early diagnosis and early treatment of PD patients are particularly important.

The clinical manifestations of Parkinson's disease include motor symptoms and non-motor symptoms (NMS), the latter of which is often ignored by clinicians. It includes common neuropsychiatric symptoms: such as depression, anxiety, apathy, lack of affect, distraction, and even hallucinations, delusions, delusions, dementia, obsessive-compulsive symptoms, panic attacks; sleep disorders: periodic limb movement disorders, excessive sleep during the day and so on. Some of these symptoms can appear before the movement disorder of Parkinson's disease, some are accompanied by the movement disorder, and some appear in the middle and late stages of Parkinson's disease, and aggravate with the aggravation of the movement symptoms. And its NMS is closely related to the severity of the entire disease of PD.

[Objective] To explore the significance of tremor analysis in judging the early diagnosis of Parkinson's disease.

Discuss the significance of tremor analysis for the prognosis of the disease. To explore the diagnostic significance of tremor analysis in patients with Parkinson's disease and benign tremor.

[Design] This is a longitudinal study to evaluate the brainstem of patients at different stages through VEMP neck, masticatory muscle and eye tests on patients with early and middle-advanced PD (20 cases each) and healthy controls (40 cases) The function of various parts is affected. At the same time, combining the patient's neurological function score and non-motor symptom score to find evidence of early involvement and early intervention.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment criteria: All patients from the outpatient and inpatient department of neurological movement disorders, aged 45-75 years, meet the following symptom scores greater than or equal to 4 points: olfactory disorder (2 points), rapid eye movement sleep behavior disorder (2 points) , Constipation (1 point), anxiety and depression symptoms (1 point), muscle stiffness (1 point), tremor (1 point), balance disorder (1 point), signed informed consent;

Exclusion Criteria:

* exclusion criteria: a. Clear cerebellar abnormalities; b. Downward vertical supranuclear gaze palsy, or selective downward vertical saccade slowed down; c. Within the first 5 years of onset, diagnosed as possible behavioral variant frontotemporal dementia or primary Progressive aphasia; d. The onset of Parkinson's syndrome that is still limited to the lower limbs for 3 years; e. Parkinson's syndrome caused by drugs; f. The effect of levodopa is not good; g. Cortical sensory loss.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parkinson's disease, the second most common neurodegenerative disease, affects 1 to 2 percent of patients over 65 years of age. China currently has nearly 2 million patients with Parkinson's disease, and the number is expected to grow exponentially in the coming years. The clinical manifestations of Parkinson's disease include tremor, rigidity, bradykinesia, postural instability and other motor symptoms. The static tremor is caused by cerebellum and basal ganglia circuits, which has nothing to do with the number of dopamine neurons. Treatment with Mdopa can reduce the tremor amplitude of patients, but generally does not change the tremor frequency.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
nigrostriatal echogenic area | 1 week after enrollment
  using the Transcranial parenchymal color Doppler ultrasound (TCS) to trace the nigrostriatal echogenic area
Electromyography (EMG) tremor analysis | 1 week after enrollment
  EMG frequency
Electromyography (EMG) tremor analysis | 1 week after enrollment
  EMG amplitude (amplitude)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoxuan Liu, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No